CLINICAL TRIAL: NCT04769011
Title: Motor Impairments in Children With Autism Spectrum Disorder: a Multimodal Approach
Acronym: MOSAICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 510
Record Dates: First submitted 2021-02-11; First posted 2021-02-24 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder; Intellectual Disability
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Intellectual Disability | interventions — Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical, neuropsychological, neurophysiological, and genetic evaluations (Experimental): Clinical, neuropsychological, neurophysiological, and genetic evaluations
  Interventions: Diagnostic Test: Clinical evaluation; Diagnostic Test: Neuropsychological evaluation; Diagnostic Test: Neurophysiological evaluation; Diagnostic Test: Genetic evaluation

INTERVENTIONS:
Diagnostic Test: Clinical evaluation — Clinical evaluation of participants by means of Autism Diagnostic Observation Schedule, Social Responsiveness Scale, Children Behavior Check List, Conners' Scale
Diagnostic Test: Neuropsychological evaluation — The participants' motor skills are measured using the Movement Assessment Battery for Children 2 (MABC2) (Henderson et al., 2007), the Developmental Coordination Disorder Questionnaire (DCDQ) (Wilson et al., 2007), and the kinematic analysis of a reach-to-drop task (Forti et al., 2011; Crippa et al., 2015).Sensorimotor domain will be also further investigated with NEPSY-II (Korkman et al., 2007) (Fingertip Tapping, Imitating Hand Positions, Manual Motor Sequences, and Visuomotor Precision).
Diagnostic Test: Neurophysiological evaluation — Magnetic Resonance Imaging (structural MRI and DTI)
Diagnostic Test: Genetic evaluation — Either blood or saliva will be obtained for participants for DNA collection. DNA will be extracted in the Molecular Biology Laboratory at the Scientific Institute IRCCS Medea. Captured exome libraries will be sequenced using the Illumina NextSeq 500 in 100 bp paired end reads. Postsequencing reads will be aligned using BWA Enrichment application on BaseSpace. VCF file will be then marked using wANNOVAR (Wang Genomics Lab). The analysis will be focused on non-synonymous variants enrichment in Gene Ontology and Human Phenotype.

SUMMARY:
The general goal of the present proposal, Progetto MOSAICO, is the identification of a multimodal panel of neuropsychological, kinematic, neurophysiological, and genetic markers associated with motor abnormalities present in ASD.

ELIGIBILITY:
Inclusion Criteria:

* having a clinical diagnosis of neurodevelopmental disorders (either ASD, ADHD, or intellectual disability) according to DSM-5 criteria;
* children with typical development are also recruited from the general population by local pediatricians or from kindergartens/schools sited near our institute

Exclusion Criteria:

* using any stimulant or non-stimulant medication affecting the central nervous system
* having an identified genetic disorder
* having vision or hearing problems
* suffering from chronic or acute medical illness.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Movement Assessment Battery for Children 2 (MABC2) | immediately after the intervention
  The MABC2 (Henderson et al., 2007) is one of the most commonly used tests for the identification of motor difficulties in children aged 3-16 years. The MABC2 includes eight subtests grouped into three areas related to different components of motor domain: manual dexterity, ball skills (such as aiming and catching), and static and dynamic balance.
Developmental Coordination Disorder Questionnaire (DCDQ) | immediately after the intervention
  The DCDQ (Wilson et al., 2007) is a parent questionnaire originally developed for estimating gross and fine motor skill difficulties in children. The questionnaire consists of 15 items investigating different subdomains of motor abilities, such as ball skills, complex motor coordination, fine and general motor skills. For each item, parents rate the children's degree of motor coordination on a 5-point scale comparing it to same-age peers.
kinematic analysis of a reach-to-drop task | immediately after the intervention
  3D kinematic data of a reach-to-drop movement are collected by a motion-capture system (The SMART D from BTS Bioengineering® - Garbagnate Milanese, Italy). The reach-to-drop task consists in reaching and grasping a ball placed over a support and dropping it in a hole (Fig. 1; Forti et al., 2011; Crippa et al., 2015). The task is simple enough to warrant compliance by all children across groups. Each participant is asked to complete at least five trials of the task with their dominant hand. Kinematic data are recorded by eight infrared-motion analysis cameras at 60 Hz with a spatial accuracy of 0.2 mm.
Magnetic Resonance (MRI) | immediately after the intervention
  Magnetic Resonance (MRI) of the Brain - MRI signal allowing tridimensional multiplanar reconstruction of the brain's structures. Anatomical images obtained with high definition T1 weighted sequences of radio frequencies - the measure is a "signal (in Hz) to noise ratio" which is obtained from each voxel (tiny 3D portions of the brain)
Diffusion Tensor Imaging (DTI) | immediately after the intervention
  Diffusion Tensor Imaging (DTI) measures of the brain microstructure and connectivity - as in all MRI techniques, the measure is a "signal (in Hz) to noise ratio" which is obtained from each voxel
Exome sequencing | immediately after the intervention
  Exome libraries will be sequenced using the Illumina NextSeq 500 in 100 bp paired end reads. Postsequencing reads will be aligned using BWA Enrichment application on BaseSpace. VCF file will be then marked using wANNOVAR (Wang Genomics Lab).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No